CLINICAL TRIAL: NCT00493142
Title: Impact of a Pre-operative Rehabilitation Exercise Program for Patients With Severe Dysfunction Awaiting Total Knee Arthroplasty
Brief Title: Pre-operative Rehabilitation Exercise Program for Total Knee Arthroplasty
Acronym: PREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Heritage Foundation for Medical Research (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-060605
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Usual care
  Interventions: Other: Usual care
- Exercise (Experimental): Exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise
  Arms: Exercise
Other: Usual care
  Arms: Usual care

SUMMARY:
The purpose of this study is to determine whether a pre-operative home rehabilitation exercise program designed for knee replacements is more effective than pre-operative usual care.

DETAILED DESCRIPTION:
Patients with lower levels of function prior to total knee arthroplasty (TKA) attain lower functional endpoints after surgery. Therapeutic exercise improves function in patients with arthritis of the knee, yet little evidence has examined the impact of pre-operative exercise for TKA.

Single blinded randomized clinical trial comparing a pre-operative home exercise program to pre-operative usual care for patients who are waiting for TKA.Comparison group is usual care within the health region which does not include pre-operative rehabilitation program.

Primary outcome: WOMAC function subscale. Secondary outcomes: 1) quality of life; 2) ambulation; 3) self-efficacy; 4) anxiety; 5) patient satisfaction; 6) cost-effectiveness of this intervention.

Total Enrollment: 230 patients

If the intervention improves function prior to surgery, results will be clinically applicable for patients waiting for surgery

ELIGIBILITY:
Inclusion Criteria:

* primary unilateral total knee arthroplasty
* poor functional status (WOMAC=50 or greater)
* 50 yrs or older
* reside within health region
* understands English

Exclusion Criteria:

* unicompartmental total knee arthroplasty
* revision surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-07; Primary Completion 2013-07 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Self-reported function | 5 evaluations within 6 months after surgery
  Self-reported function

SECONDARY OUTCOMES:
Quality of life, self-efficacy, ambulation, anxiety and patient satisfaction | 5 evaluations within 6 months after surgery
  Quality of life
self-efficacy | 5 evaluations within 6 months after surgery
  self-efficacy
ambulation, anxiety and patient satisfaction | 5 evaluations within 6 months after surgery
  ambulation
anxiety | 5 evaluations within 6 months after surgery
  anxiety
patient satisfaction | 5 evaluations within 6 months after surgery
  patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Allyson Jones, PhD, Principal Investigator — University of Alberta; Lauren Beaupre, PhD, Study Director — Capital Health- UAH
Locations (1):
- University of Alberta- Capital Health, Edmonton, Alberta, Canada